CLINICAL TRIAL: NCT07240584
Title: The Impact of Exercise Prehabilitation on Upper Extremity Range of Motions, Functionality and Quality of Life in Breast Cancer Survivors: A Prospective Clinical Trial
Brief Title: Exercise Prehabilitation of Breast Cancer
Acronym: Prehab of BC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Balikesir Hospital Eduation and Research (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UHS Balikesir H PMR
Record Dates: First submitted 2025-11-16; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Shoulder Dysfunction; Quality of Life; Postoperative Recovery; Fatigue; Lymphedema
Keywords: exercise prehabilitation; breast cancer; upper extremity functionality; quality of life
MeSH Terms: conditions — Breast Neoplasms; Fatigue; Lymphedema

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group Assignment (Other)
  Interventions: Behavioral: Exercise-Based Prehabilitation Program

INTERVENTIONS:
Behavioral: Exercise-Based Prehabilitation Program — The exercise program was delivered to patients through both visual and written materials, accompanied by face-to-face training sessions conducted by a physiotherapist. A home-based program was designed separately for the pre-surgery phase, postoperative day 1, day 3, day 7, and the maintenance period.
  The exercise template included postural correction, breathing, aerobic, stretching, and resistive strengthening exercises targeting muscles in adjacent to the shoulder joint and mobilization of scapulothoracic complex via stretching and strengthening exercises of periscapular muscles.

SUMMARY:
This prospective prehabilitation trial evaluated the effectiveness of an individualized exercise program initiated before breast cancer surgery and maintained for 12 months. The intervention aimed to promote functional recovery and improve patient-reported outcomes.

DETAILED DESCRIPTION:
Women scheduled for breast surgery due to breast cancer were enrolled in an individualized prehabilitation program that began in the preoperative period and continued for 12 months. The exercise program included range-of-motion, strengthening, and postural correction exercises delivered through supervised and home-based sessions. Outcomes were evaluated at baseline and at 1st, 3rd, 6th, and 12th months. Functional outcomes, shoulder range of motion, pain intensity, lymphedema development, and patient-reported quality of life were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Female patients diagnosed with breast cancer scheduled for surgical treatment
* Age ≥ 18 years
* Able to perform exercise
* Provided informed consent

Exclusion Criteria:

* Metastatic disease
* Prior upper limb injury or neurologic impairment
* Inability to comply with exercise program
* Postoperative chemotherapy before the 3rd month

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 30 (Actual)
Dates: Start 2024-10-25 (Actual); Primary Completion 2025-11-02 (Actual); Study Completion 2025-11-02 (Actual)

PRIMARY OUTCOMES:
Shoulder Range of Motion | baseline, 1st-3rd-6th-12th month
  Measurement of Flexion, Abduction, Internal and External Rotation of Shoulder with goniometer
Pain Intensity | baseline, 1st-3rd-6th-12th month
  measure of pain with VAS (Visual analog scale)
Functional Outcomes | baseline and 12th month
  measure of upper extremity functions with UEFI-15 (Upper extremity functional index) instrument

SECONDARY OUTCOMES:
fatigue | baseline and 12th month
  measure of fatigue condition with FSS (Fatigue severity scale) instrument
Quality of Life impairment | baseline and 12th month
  measure of Quality of Life with EORTC-QLQ-C30 (European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire) instrument
lymphedema | baseline and 12th month
  Limb volume difference >10% or clinical signs of edema

CONTACTS AND LOCATIONS:
Locations (1):
- Balikesir Ataturk City Hospital Affiliated with University of Health Sciences, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Brahmbhatt P, Sabiston CM, Lopez C, Chang E, Goodman J, Jones J, McCready D, Randall I, Rotstein S, Santa Mina D. Feasibility of Prehabilitation Prior to Breast Cancer Surgery: A Mixed-Methods Study. Front Oncol. 2020 Sep 25;10:571091. doi: 10.3389/fonc.2020.571091. eCollection 2020. PMID 33072603
- [Result] Michael CM, Lehrer EJ, Schmitz KH, Zaorsky NG. Prehabilitation exercise therapy for cancer: A systematic review and meta-analysis. Cancer Med. 2021 Jul;10(13):4195-4205. doi: 10.1002/cam4.4021. Epub 2021 Jun 10. PMID 34110101
- [Result] Alicia DRJ, Manuel GS, Ignacio CVA. Physical prehabilitation in patients with breast cancer: a systematic review. Support Care Cancer. 2025 Jan 6;33(1):71. doi: 10.1007/s00520-024-09122-w. PMID 39757306